CLINICAL TRIAL: NCT05853107
Title: Pilot Study of AuTNA I (Au Nanoparticle-decorated TiO2 Nanowire Arrays, Retinal Prothesis) -a Safety and Efficacy Evaluation.
Brief Title: Pilot Study of AuTNA I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AuTNA I
Record Dates: First submitted 2023-04-15; First posted 2023-05-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant AuTNA I (Experimental): This is a single arm study where the status and performance of the implanted eye prior to the surgery serves as the comparator.
  Interventions: Device: AuTNA I

INTERVENTIONS:
Device: AuTNA I — AuTNA I means Au nanoparticle-decorated TiO2 Nanowire Arrays, a retinal prothesis designed for subretinal implantation.

SUMMARY:
The objective of the study is to evaluate:

1. Safety of AuTNA I for subretinal implantation in patients with retinitis pigmentosa;
2. Efficacy of AuTNA I for subretinal implantation in patients with retinitis pigmentosa.

DETAILED DESCRIPTION:
In this study, AuTNA I (nanoparticle-decorated TiO2 Nanowire Arrays), which is designed to replace the damaged photoreceptors in RP patients, was implanted in one eye of the subjects. The change or improvement in the visual acuity of the subjects, as well as the potential side effects, was then fully evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years of age.
2. Clinically diagnosed as retinitis pigmentosa (one of the following two conditions):

   ① typical triadfundus manifestations: "osteoblastic" pigmentation of retina, arterial stenosis, and waxy atrophy of optic disc.

   ② typical fundus changes with both a and b, with or without c:
   1. poor night vision before vision loss;
   2. standard 5 ERG examination showing more severely damaged scotopic response than photopic, even non response
   3. impaired peripheral visual field in perimetry (when the patient's vision permits).
3. No or suspicious light perception in the eye for AuTNA I implantation.
4. Intact inner retinal structure on OCT. No macular retinal or choroidal neovascularization.
5. Voluntary to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Entities that might interfere with the functioning of AuTNA I, e.g. open ocular trauma, retinal detachment, glaucoma, severe uveitis, etc.
2. Uncontrolled systemic diseases including hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg), diabetes (blood glucose ≥8.0mmol/L with medication);
3. Allergic constitution.
4. Entities that might prevent the observation of the fundus, e.g. corneal opacity, etc.
5. Ocular disease not suitable for undertaking the implantation surgery, e.g. corneal ulcers, etc.
6. Habits of rubbing the eyes.
7. Compromised liver function (ALT and AST 1.5 times over the normal limits), renal function (Cr 1.5 times over the normal limits), coagulation function (APTT 1.5 times over the normal limits).
8. Pregnancy, lactating or planning to be pregnant within 6 months.
9. History of epilepsy or serious psychiatric diseases.
10. Other local or systemic diseases that may affect the vision.
11. Participation in other clinical trials within 1 month before this study.
12. Other conditions that the researcher found imporper to be included into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
FST | Baseline and improvement of FST at 3 months.
  FST means Full-field Sensitivity Threshold. The thresholds of light with different wavelengths. The exam was performed at baseline and at various time points throughout the first year after the implantation.
BCVA | Baseline and improvement of BCVA at 3 months.
  BCVA means Best-Corrected Visual Acuity, and is measured by Snellen Chart, EDTRS Chart and charts designed for people with low vision. It's performed at baseline and at various timepoints throughout the first year after the implantation.
Clinical electrophysiology of vision | Baseline and improvement of electrophysiology at 3 months.
  Electrophysiological examinations of the visual pathway to evaluate the light responsiveness, including VEP, ERG and mfERG (Multifocal ERG). It's performed at baseline and at various timepoints throughout the first year after the implantation.
ElectroEncephaloGram | Baseline and change of EEG at 3 months.
  EEG(ElectroEncephaloGram) target frequency power amplitude and signal-to-noise ratio (SNR) would be used to analyse the visual stimulus steady-state evoked potential paradigms. It's performed at baseline and at various timepoints throughout the first year after the implantation.
Functional Magnetic Resonance Imaging | Baseline and change of fMRI at 3 months.
  Using fMRI (Functional Magnetic Resonance Imaging) to measure visual stimulus-induced brain activity caused by changes in blood flow. It's performed at baseline and at various timepoints throughout the first year after the implantation.

SECONDARY OUTCOMES:
Visual field | Recruitment (baseline) and 3 months, 6 months and 1 year after implantation.
  The visual sensitivity of the implantation site of the fundus is measured with microfield perimetry. It's performed at baseline and at various timepoints throughout the first year after the implantation.
Line task | Recruitment (baseline) and 3 months, 6 months and 1 year after implantation.
  To record the completion (completed/failed, time course if completed) of walking along a five-meter-long white strip on the black floor in a well-illuminated environment. It's performed at baseline and at various timepoints throughout the first year after the implantation.
VisQoL | Recruitment (baseline) and 3 months, 6 months and 1 year after implantation.
  Vision-related quality of life is assessed with the VisQoL (Vision and Quality of Life) scale. It's performed at baseline and at various timepoints throughout the first year after the implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Chunhui Jiang, Study Director — Eye and ENT Hospital of Fudan University
Locations (1):
- Chunhui Jiang, Shanghai, Shanghai Municipality, China